CLINICAL TRIAL: NCT01806389
Title: Lactation Among Buprenorphine Maintained Women: A Pilot Study
Brief Title: A Study of Breastfeeding in Buprenorphine Maintained Women
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Lauren M. Jansson, Associate Professor of Pediatrics Johns Hopkins University School of Medicine, Johns Hopkins University
Other Study IDs: NA_00080884
Record Dates: First submitted 2013-02-20; First posted 2013-03-07 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-02

CONDITIONS: Opioid Dependency
Keywords: Breast milk; Breastfeeding; Lactation; Buprenorphine; Opioid
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal urine, plasma and breast milk INnfant plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Buprenorphine: Buprenorphine maintained women at delivery of their infant

SUMMARY:
Goals: The overarching goals for this proposed research are to provide pilot data for a study to inform the FDA regarding the safety of breastfeeding infants of mothers on buprenorphine maintenance and to develop guidelines for the practitioner treating buprenorphine maintained women who wish to breastfeed.

Background: There is an increase in the prevalence of illicit opiate use among women of childbearing age. Recently, a large multisite study has suggested buprenorphine as an alternative to methadone for use in this population. As a consequence, buprenorphine is likely to be delivered to larger populations of pregnant and post-partum women. The population of prenatally opioid-exposed neonates is a particularly vulnerable population. Advances in neuroscience, molecular biology and epigenetics indicate that greater attention should be given to strategies that prevent, reduce, or mitigate the consequences of significant adversity on the developing brain. Breast milk and breastfeeding offer significant health and other benefits that are particularly salient for this group. Today, there is a near complete lack of information regarding the safety of buprenorphine maintenance and lactation, making it unlikely that providers will endorse or mothers will adopt this practice.

Methods: Five pregnant buprenorphine maintained breastfeeding women and their neonates will be enrolled. Subjects will selected by buprenorphine maintenance in the postpartum period and enrollment in a parent protocol and by decision to breast feed their infants. Subject will provide breast milk at times of peak maternal buprenorphine levels on days 2, 3, 4, 14 and 30 after delivery to determine buprenorphine and norbuprenorphine concentrations. Subjects will also provide plasma at times of peak buprenorphine levels for determination of buprenorphine and norbuprenorphine concentrations on the same days. Concentrations of buprenorphine and norbuprenorphine in the plasma of infants will be determined on approximately day 14 of life. The relationship between maternal dose, maternal and infant plasma concentrations, and breast milk concentrations of buprenorphine and norbuprenorphine will be determined, and ingestible infant dose calculated.

DETAILED DESCRIPTION:
This study recruits participants from a funded trial evaluating fetal neurobehavior and maternal physiology among a population of opioid dependent and buprenorphine maintained pregnant women. Those women electing to breastfeed will be approached for participation in this study at 36 weeks of gestation.

Study Procedures Study participants will have urine toxicology testing for the following drug classes/cut off values: cocaine/300 ng/mL; methamphetamines/1000ng/mL; methadone/300ng/mL; MDMA/500 ng/mL; MOP/300 ng/mL; oxycodone/100 ng/mL; PCP/25 ng/mL; benzodiazepines/300ng/mL; buprenorphine/10 ng/mL; marijuana/50ng/mL weekly as part of study procedures in addition to weekly random urine toxicology screening provided at CAP for the study period of 36 weeks until delivery. To ensure that participants are not using illicit substances or abusing licit substances and are candidates for the institution and continuation of breastfeeding, subjects will continue to provide urine toxicology testing as above for the period of time from delivery to day 30 postpartum. Subjects noted to be doing so will be discharged from the protocol and referred to their substance abuse treatment counselor for appropriate consequences.

Data collection protocol: Upon delivery, the nursing staff at the hospital of delivery will contact study staff for initiation of study procedures. Women will have plasma and breast milk samples obtained by study personnel on days 2, 3, 4, 14 and 30 at times of peak (2 ½ hours after sublingual dosing) maternal buprenorphine levels. Infant weight will be collected on these days. Days of data collection will be determined by the, 2nd, 3rd, 4th 24 hour periods after birth of the infant. The 14th, and 30th day data collections will occur on the weekday nearest the 24 hour period on those days. Infant NICU Network Neurobehavioral Scale scores on days 3, 14 and 30 and infant NAS scores as below are collected as part of the parent protocol and data abstracted for this protocol.

Maternal plasma: Using 3mL vacutainer green-top collection tubes, 3 cc of blood will be collected via venupuncture by one of two study RNs, one responsible for inpatient specimen collection (i.e. while the mother and infant are hospitalized after delivery) and one responsible for outpatient specimen collection (after hospital discharge). Blood samples will be collected on ice and within two hours, cold centrifuged to harvest the plasma. Plasma will be stored in polypropylene tubes and stored at -20°C. Plasma will be collected at times of peak maternal buprenorphine levels on days 2, 3, 4, 14 (approximately) and 30 (approximately) after infant delivery.

Breast milk: Breast milk samples will be collected after the infant has completed feeding from the same breast via electric pump and consist of approximately 5 cc of breast milk at time of peak maternal buprenorphine levels on days 2,3,4, 14 and 30 after infant delivery. Breast milk will be stored at -20°C within two hours of collection.

Analysis of breast milk and plasma samples: Plasma and breast milk samples will be analyzed by the Chemistry and Drug Metabolism Section of the Intramural Research Program of the National Institute on Drug Abuse, National Institutes of Health in Baltimore, Maryland under the direction of Dr. Marilyn A. Huestis.

Infant plasma: 1cc of infant blood will be taken by heel stick on the weekday nearest day 14 of life. The 14 day blood sample will be coincident with a routine infant blood test (PKU testing) when possible. Blood samples will be collected on ice and within two hours, cold centrifuged to remove plasma. Plasma will be stored in polypropylene tubes and stored at -20°C until analysis.

Other infant data: Infant weight will be obtained at each data collection point (i.e. days 2,3,4, 14 and 30).

Other maternal data: Maternal compliance to drug treatment will be abstracted from daily treatment records. Poor compliance to treatment will be determined on an individual basis via discussion with the subject's counselor, but in general compliance will be determined by attendance to daily therapy at CAP with no unexcused or unexplained absence from treatment in the 30 days subsequent to delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-41 years
2. Opioid dependent per DSMIVR criteria, buprenorphine maintained, enrolled in parent study.
3. Delivery at 37 weeks of gestation or later
4. Breast feeding in the first month of life

Exclusion Criteria:

1. Concurrent Axis I diagnosis, or the presence of a serious psychiatric illness that would preclude informed consent
2. Major congenital malformation or minor congenital malformation that would impair the infant's ability to feed (i.e. Pierre-Robin syndrome, cleft palate)
3. Delivery at an outside institution unaffiliated with this protocol
4. Failure to leave specimens as per protocol
5. Infant medical complications that impair the ability to feed after delivery (i.e. respiratory concerns such as meconium aspiration, perinatal asphyxia, etc. These will be individually determined on a case-by-case basis)
6. Any detected maternal medical condition making lactation inadvisable, i.e. newly diagnosed HIV infection or requirement for medication not compatible with breastfeeding.
7. Infants with other medical conditions that would make study participation impossible, i.e. nonviable neonates, neonates with uncertain viability.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ten buprenorphine maintained women who deliver and infant and desire to breastfeed
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Jansson, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jansson LM, Spencer N, McConnell K, Velez M, Tuten M, Harrow CA, Jones HE, Swortwood MJ, Barnes AJ, Scheidweiler KB, Huestis MA. Maternal Buprenorphine Maintenance and Lactation. J Hum Lact. 2016 Nov;32(4):675-681. doi: 10.1177/0890334416663198. Epub 2016 Sep 26. PMID 27563013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a study evaluating fetal and infant effects of maternal buprenorphine treatment
Pre-assignment Details: Fourteen women were consented for this protocol but 4 were withdrawn for various reasons, i.e. inability to provide samples, changed mind about breastfeeding.
Groups:
- Buprenorphine Maintained Lactating Women: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria
Period: Overall Study
Arm/Group | Buprenorphine Maintained Lactating Women
Started | 14
Completed | 10
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Buprenorphine Maintained Lactating Women
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maternal Plasma Concentrations of Buprenorphine
Description: Maternal plasma will be obtained at the time of peak buprenorphine levels on days 2,3,4,14 and 30
Time Frame: Days 2,3,4,14 and 30 after delivery
Measure: Median (Full Range); unit: ug/mL
Groups:
- PLASMA Buprenorphine Maintained Lactating Women Day 2: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing plasma for analysis on day 2
- PLASMA Buprenorphine Maintained Lactating Women Day 3: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing plasma for analysis on day 3
- PLASMA Buprenorphine Maintained Lactating Women Day 4: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing plasma for analysis on day 4
- PLASMA Buprenorphine Maintained Lactating Women Day 14: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing plasma for analysis on day 14
- PLASMA Buprenorphine Maintained Lactating Women Day 30: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing plasma for analysis on day 30
Arm/Group | PLASMA Buprenorphine Maintained Lactating Women Day 2 | PLASMA Buprenorphine Maintained Lactating Women Day 3 | PLASMA Buprenorphine Maintained Lactating Women Day 4 | PLASMA Buprenorphine Maintained Lactating Women Day 14 | PLASMA Buprenorphine Maintained Lactating Women Day 30
Number analyzed (Participants) | 10 | 10 | 9 | 9 | 8
ug/mL | 1.2 [0.4 to 6.1] | 1.7 [0.7 to 7.0] | 2.0 [0.5 to 5.9] | 2.4 [0.7 to 3.3] | 2.2 [1.2 to 6.1]

2. Primary Outcome: Maternal Breast Milk Concentrations of Buprenorphine
Description: Breast milk will be obtained on these days at the time of peak plasma levels of buprenoprhine
Time Frame: Days 2,3,4,14 and 30 after delivery
Measure: Median (Full Range); unit: ug/mL
Groups:
- BREAST MILK Buprenorphine Maintained Lactating Women Day 2: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing breast milk for analysis on day 2
- BREAST MILK Buprenorphine Maintained Lactating Women Day 3: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing BREAST MILK for analysis on day 3
- BREAST MILK Buprenorphine Maintained Lactating Women Day 4: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing BREAST MILK for analysis on day 4
- BREAST MILK Buprenorphine Maintained Lactating Women Day 14: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing BREAST MILK for analysis on day 14
- BREAST MILK Buprenorphine Maintained Lactating Women Day 30: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing BREAST MILK for analysis on day 30
Arm/Group | BREAST MILK Buprenorphine Maintained Lactating Women Day 2 | BREAST MILK Buprenorphine Maintained Lactating Women Day 3 | BREAST MILK Buprenorphine Maintained Lactating Women Day 4 | BREAST MILK Buprenorphine Maintained Lactating Women Day 14 | BREAST MILK Buprenorphine Maintained Lactating Women Day 30
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 7
ug/mL | 2.3 [0.2 to 4.2] | 1.5 [0.2 to 5.0] | 1.4 [0.3 to 5.2] | 4.8 [1.0 to 10.5] | 3.3 [2.2 to 20.8]

3. Primary Outcome: Infant Plasma Concentrations of Buprenorphine
Description: Infant plasma concentrations of buprenoprhine obtained on day 14 of life
Time Frame: Day 14 of life
Measure: Median (Full Range); unit: ug/mL
Groups:
- INFANT PLASMA Buprenorphine Maintained Lactating Women Day 14: Buprenorphine maintained women at delivery of their infant opting to breastfeed their infants and meeting study criteria and providing INFANT PLASMA for analysis on day 14
Arm/Group | INFANT PLASMA Buprenorphine Maintained Lactating Women Day 14
Number analyzed (Participants) | 9
ug/mL | 0 [0 to 2.9]

ADVERSE EVENTS:
Arm/Group | Buprenorphine
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Small group size Variable amounts of breast milk received by the majority of the sample Reports of exclusive breastfeeding vs formula supplementation were by maternal report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No